CLINICAL TRIAL: NCT03977051
Title: Exploring Immunosuppressant Medication Adherence in Kidney Transplant Patients
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 16HH3697
Record Dates: First submitted 2017-04-25; First posted 2019-06-06 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Adherence, Medication; Transplantation, Kidney
Keywords: Kidney transplantation
MeSH Terms: conditions — Medication Adherence | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focus group: Focus group to explore immunosuppressant medication adherence in kidney transplant patients
  Interventions: Behavioral: Focus group

INTERVENTIONS:
Behavioral: Focus group — Kidneys transplant patients will discuss their attitudes and beliefs towards immunosuppressant medication adherence

SUMMARY:
To describe the beliefs, understanding and experience of immunosuppressant medication adherence in our current transplant patient population through a series of patient focus groups

DETAILED DESCRIPTION:
The investigators want to understand more about why some of our kidney transplant patients find it difficult to take their anti-rejection medicines as intended. It is hoped that if the investigators can improve their understanding of why some patients struggle with their anti-rejection medicines, the investigators will be able to find better ways to help our transplant patients and so fewer patients may develop problems with their transplant. This study will collect qualitative data from a series of focus groups with kidney transplant recipients to explore their beliefs, understanding and experience of anti-rejection medication adherence. The focus groups will also explore the support that participants have received to help them with their medication adherence and what support they feel should be available to them and to others in the future to optimise anti-rejection medication adherence in transplant patients. Five focus groups will be undertaken. Each focus group will include six patients and will last for approximately 1.5 hours. All participants will be kidney transplant recipients transplanted and followed up at Imperial College Renal and Transplant Centre.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients transplanted and under the active follow up of ICRTC.
* Speak and understand English
* 18 years and above

Exclusion Criteria:

* Unable to speak and understand English
* Below 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Goodall, MSC, BSc, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Renal and Transplant Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Focus Group
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Focus Group
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: years] | 56.19 [26.53 to 72.33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 4
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 26
Years since transplant [Mean (Full Range); unit: years] | 4.35 [0.19 to 13.99]

OUTCOME MEASURES:

1. Primary Outcome: Number of Kidney Transplant Patients Who Expressed an Understanding of the Term Immunosuppression Medication Adherence and the Importance Immunosuppression Medication Adherence Post Transplant
Description: Through a series of focus groups, the investigators will qualitatively explore kidney transplant patients' understanding of the terms immunosuppressant medication adherence and nonadherence. What importance do patients attach to adherence. Do patients understand that nonadherence may effect the outcome of the transplant. The focus groups will identify the common practical and perceptual barriers to adherence identified by transplant patients and the interventions kidney transplant patients have used to try and improve their adherence. The focus groups will identify which interventions patients have found effective and which interventions patients have not found to be effective to improve their adherence. They will also identify support patients have had with adherence since their transplant, the support patients feel could have helped them to better adhere to their medicines up to now and the support our patients feel would help them to adhere better to their medicines in the future
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Focus Group
Number analyzed (Participants) | 26
Participants
  Good understaning of the term | 19
  Good understanding risk of rejection / graft loss | 19

2. Primary Outcome: Number of Kidney Transplant Patients Who Identified Interventions to Support Immunosuppressant Medication Adherence
Description: as for outcome 1
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Focus Group
Number analyzed (Participants) | 26
Participants
  Medicines compliance aids, smart-phone apps | 14
  Support provided to them by the MDT | 26
  Use of alarms and apps | 15

3. Primary Outcome: Number of Patients Who Identify Barriers to Immunosuppression Medication Adherence
Description: as for outcome 1
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Focus Group
Number analyzed (Participants) | 26
Participants
  Forgetfulness / recall | 6
  Ability to take at regular time / on emtpy stomach | 6
  Adverse effects | 1

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Focus Group
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT03977051/Prot_SAP_000.pdf